CLINICAL TRIAL: NCT06407713
Title: Effects of Intrinsic Foot Muscle Training With and Without Hip Abductor Muscle Strengthening on Pain and Functional Mobility in Patients With Pronation Distortion Syndrome
Brief Title: Intrinsic Foot Muscle Training With and Without Hip Abductor Muscle Strengthening in Pronation Distortion Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0186
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Pronation Deformity of the Foot
Keywords: Exercise; Functional Mobility; Muscle strength; Navicular drop; Pain; Pronation
MeSH Terms: conditions — Motor Activity; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intrinsic foot muscle training. (Active Comparator): Intrinsic foot muscle training would be performed
  Interventions: Other: Intrinsic foot muscle training
- intrinsic foot muscle training with hip abductor muscle training (Active Comparator): hip abductor muscle strengthening would be administered alongside intrinsic foot muscle training
  Interventions: Other: Intrinsic foot muscle training; Other: Hip abductor muscle training

INTERVENTIONS:
Other: Intrinsic foot muscle training — The duration of intervention will be 6 weeks, 3 sessions a week, a total of 18 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with intrinsic foot muscle training
Other: Hip abductor muscle training — The duration of intervention will be 6 weeks, 3 sessions a week, a total of 18 sessions will be given to the study participants. Each session will last for 30 minutes. Conventional physical therapy will be given to participants along with hip abductor muscle training
  Arms: intrinsic foot muscle training with hip abductor muscle training

SUMMARY:
Pronation distortion syndrome is one of the most common abnormalities in the lower extremity that causes alterations in the structures of the skeletal parts of the foot. The aim of the study will be to compare the effects of intrinsic foot muscle with and without hip abductor muscle strengthening on pain and functional mobility in patients with Pronation Distortion Syndrome.

DETAILED DESCRIPTION:
A Randomized Clinical Trial will be conducted at Nawaz Sharif Social Security Hospital, Multan Road, Lahore through convenience sampling technique on 54 patients which will be allocated using simple random sampling through computer generated method into Group A and Group B. Group A will be treated with intrinsic foot muscle training at the frequency of 4 sets with 15 repetitions and Group B will be treated with hip abductor muscle strengthening at the frequency of 3 sets with 15 repetitions; session would be conducted thrice a week. Outcome measures will be conducted through numeric pain scale and lower extremity functional scale after 6 weeks. Data will be analyzed during SPSS software version 25. After assessing normality of data by Kolmogorov-Smirnov test, it will be decided either parametric or non-parametric test will be used within a group or between two groups.

ELIGIBILITY:
Inclusion Criteria:

* Ages 20-30 years
* Both male and female gender
* Foot pronation on observation
* Navicular Drop Test more than 10 mm (measured in weight bearing and non- weight bearing positions distance between ground and navicular tuberosity and difference calculated)
* Increased Q angle : Males: > 16; females >18

Exclusion Criteria:

* Other deformities such as tarsal coalition and vertical talus
* Any history of surgery involving both lower extremities
* Neuromuscular disorder

Ages: 20 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2024-05-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-08-15 (Actual)

PRIMARY OUTCOMES:
NPRS | 6th week
  Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain Changes from base Line Numeric Pain rating scale is a scale for pain starting from 0-10. where 0 indicate no pain and 10 indicate severe pain The Numerical Pain Rating Scale (NPRS) is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain).
Navicular drop test | 1st day
  Used as an indicator of foot. Height of the navicular tuberosity from the ground is measured with the subject being non-weight bearing and then weight bearing, height of the navicular tuberosity is measured. The difference is determined. A difference of 10 > mm will be considered as flexible flatfoot. ND test has proven valid and reliable for the assessment of the medial arch
Lower extremity functional scale | 6th week
  The Lower Extremity Functional Scale (LEFS) is a questionnaire containing 20 questions about a person's ability to perform everyday tasks. The LEFS can be used by clinicians as a measure of patients' initial function, ongoing progress and outcome, as well as to set functional goals. It will be used to monitor the patient over time and to evaluate the effectiveness of the interventions.
Universal goniometer | 6th week
  Universal goniometer is a tool that measures an angle or permits the rotation of an object to a definite position. It- has three parts: body, fulcrum and arms (stationary and moving)

CONTACTS AND LOCATIONS:
Overall Officials: Rabiya Noor, PHD, Principal Investigator — Study Principal Investigator
Locations (1):
- Nawaz Sharif social security hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mulligan EP, Cook PG. Effect of plantar intrinsic muscle training on medial longitudinal arch morphology and dynamic function. Man Ther. 2013 Oct;18(5):425-30. doi: 10.1016/j.math.2013.02.007. Epub 2013 Apr 28. PMID 23632367
- [Background] Elsayed W, Alotaibi S, Shaheen A, Farouk M, Farrag A. The combined effect of short foot exercises and orthosis in symptomatic flexible flatfoot: a randomized controlled trial. Eur J Phys Rehabil Med. 2023 Jun;59(3):396-405. doi: 10.23736/S1973-9087.23.07846-2. Epub 2023 Mar 29. PMID 36988565
- [Background] Lee DR, Choi YE. Effects of a 6-week intrinsic foot muscle exercise program on the functions of intrinsic foot muscle and dynamic balance in patients with chronic ankle instability. J Exerc Rehabil. 2019 Oct 28;15(5):709-714. doi: 10.12965/jer.1938488.244. eCollection 2019 Oct. PMID 31723561
- [Background] Kim JS, Lee MY. The effect of short foot exercise using visual feedback on the balance and accuracy of knee joint movement in subjects with flexible flatfoot. Medicine (Baltimore). 2020 Mar;99(13):e19260. doi: 10.1097/MD.0000000000019260. PMID 32221061
- [Background] Pabon-Carrasco M, Castro-Mendez A, Vilar-Palomo S, Jimenez-Cebrian AM, Garcia-Paya I, Palomo-Toucedo IC. Randomized Clinical Trial: The Effect of Exercise of the Intrinsic Muscle on Foot Pronation. Int J Environ Res Public Health. 2020 Jul 7;17(13):4882. doi: 10.3390/ijerph17134882. PMID 32645830